CLINICAL TRIAL: NCT05008302
Title: Age and Body Position on Handgrip Strength and Movement Coordination of Upper Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Olczak (Other)
Responsible Party: Sponsor-Investigator, Anna Olczak, PhD; Senior Specjalit of the Rehabilitation Clinc, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2/KRN/2019
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Stroke
Keywords: stroke; age; grip strength; coordination movement; stabilization
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To improve the coordination of the wrist and hand after stroke in three age groups. (Experimental): The test consisted of two motor tasks, carried out in two different starting positions: sitting and lying down (supine). During the first examination, the subject sat on the therapeutic table (without back support), feet resting on the floor. The upper limb was to be examined in adduction, with the elbow bent in the intermediate position between pronation and supination of the forearm. In the supine position, the upper limb was stabilized at the subject's body (adduction in the humeral joint, elbow flexion in the intermediate position).
  Interventions: Procedure: hand motor coordination in a sitting positin

INTERVENTIONS:
Procedure: hand motor coordination in a sitting positin — Before each test, the patient was instructed on how the exercise should be done. The test consisted of two motor tasks, carried out in two different starting positions: sitting and lying down (supine). During the first examination, the subject sat on the therapeutic table (without back support), feet resting on the floor. The upper limb was to be examined in adduction, with the elbow bent in the intermediate position between pronation and supination of the forearm. In the supine position, the upper limb was stabilized at the subject's body (adduction in the humeral joint, elbow flexion in the intermediate position).
  Other Names: hand motor coordination in a supine position

SUMMARY:
The aim of the study was to analyze the importance of the position of the body and the examined upper limb on the parameters of movement coordination and hand grip strength in various age groups of people after a stroke and healthy individuals.

DETAILED DESCRIPTION:
The aim of this experiment was to analyze the parameters of motor coordination and handshake strength in stroke patients and healthy volunteers in various age groups and selected torso and upper limb positions. Both patients and healthy volunteers were prospectively divided into three age groups: 18-45, 46-60 and 61 and above. Thus, the maximum range of motion (ROM), frequency of wrist and finger movements, and grip strength (dependent variables) were valued in three age groups and different starting positions (independent variables). The Hand Tutor device (MediTouch, Israel) and the electronic manual dynamometer EH 101 (Camry, China) for grip strength measurement (error of measurement, 0.5 kg/lb) were used.

The Hand Tutor allows measurements of the frequency of movement (i.e., the number of cycles per second, where one cycle represents the movement from flexion to contraction) and the maximum range of movement, which is automatically measured during the frequency test, were performed over time 10 seconds (sensitivity: 0,05 [mm] of wrist and fingers Ext./Flex), the frequency of movement (motion capture speed: up to 1 [m/sec]).

The test consisted of two motor tasks, carried out in two different starting positions: sitting and lying down (supine). During the first examination, the subject sat on the therapeutic table (without back support), feet resting on the floor. The upper limb was to be examined in adduction, with the elbow bent in the intermediate position between pronation and supination of the forearm. In the supine position, the upper limb was stabilized at the subject's body (adduction in the humeral joint, elbow flexion in the intermediate position).

In each of the starting positions, after putting the glove on, the subject was asked to make moves as quickly and in as full a range as possible. Finally, the measurement of grip strength with a dynamometer was performed in both analyzed starting positions, after completing the range of motion and speed or frequency tests. The upper extremity tested in stroke patients was the paretic extremity. In healthy subjects, the dominant hand was tested.

ELIGIBILITY:
Inclusion Criteria:1) patients with ischemic stroke; 2) Trunk Control Test 70-100 points; 3) subjects who were in a state allowing movements of the upper extremity (FMA-UE 40-66 motor function points); 4) muscle tension (MAS 0 -1+); 5) no severe deficits in communication, memory, or understanding; 6) at least 18 years of age.

-

Exclusion Criteria:1) stroke up to four weeks after the episode, 2) another neurological disease entity 3) lack of trunk stability, 4) no wrist and hand movement, 5) muscle tension (˃2 MAS), 6) high or very low blood pressure, 7) severe deficits in communication, memory, or understanding; dizziness, the malaise of the respondents.

Control group inclusion criteria: 1) the control group consisted of healthy subjects, free from the upper extremity motor coordination disorders; 2) at least 18 years of age.

Control group exclusion criteria: 1) a history of neurologic or musculoskeletal disorders such as carpal tunnel syndrome, tendonitis, stroke, head injury, or other conditions that could affect their ability to active movement and grip hand; 2) severe deficits in communication, memory, or understanding.

-

Ages: 22 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Maximum range of movement of the wrist [mm] | up to 1 week
  Hand Tutor allows measurements of the maximum range of motion (ROM).
Frequency of wrist movement (flexion to extension), cycles#/sec | up to 1 week
  The Hand Tutor allows measurements the speed or frequency (i.e., the number of cycles
Frequency of 1st, 2nd, 3rd, 4th, 5th finger movement (flexion to extension), cycles#/sec | up to 1 week
  The Hand Tutor allows measurements the speed or frequency (i.e., the number of cycles
1st, 2nd, 3rd, 4th, 5th finger maximum range of motion (ROM), [mm] | up to 1 week
  The Hand Tutor allows measurements of the maximum range of motion (ROM).
Assessment of the grip strength | up to 1 week
  Grip strength, kg (a manual electronic dynamometer (EH 101) was used for grip strength measurement (error of measurement, 0.5 kg/lb)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Olczak, PhD, Principal Investigator — Military Institute of Medicine
Locations (1):
- Anna Olczak, Warsaw, Masovian District, Poland